CLINICAL TRIAL: NCT01019772
Title: A Multicentre, Comparative, Two-arm, Parallel-group, Double-blind, Randomized Phase III Study to Assess Immunogenicity and Safety of LBVH0101 (Haemophilus Influenzae Type b Tetanus Toxoid Conjugate Vaccine) Compared With Hiberix™ Vaccine in Healthy Infants at Two, Four and Six Months of Age
Brief Title: Immunogenicity and Safety Study of LBVH0101 in Healthy Infants at Two, Four and Six Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Gyoung-Jin Choi/Assistant manager, LG Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LG-VHCL002
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Infectious Disease by Haemophilus Influenzae Type b
MeSH Terms: interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LBVH0101 (Experimental)
  Interventions: Biological: LBVH0101 (Hib vaccine)
- Hiberix (Active Comparator)
  Interventions: Biological: Hiberix™ Vaccine

INTERVENTIONS:
Biological: LBVH0101 (Hib vaccine)
  Arms: LBVH0101
Biological: Hiberix™ Vaccine
  Arms: Hiberix

SUMMARY:
The purpose of this study is to evaluate and compare the immunogenicity and safety of LBVH0101 (Haemophilus influenzae type b tetanus toxoid conjugate vaccine) to that of Hiberix™ at vaccination in healthy infants at their 2, 4, and 6 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infants aged from 49 days to 84 days at the time of enrollment.
* The gestation period was 37 weeks or longer, and birth weight was 2.5 kg or more.
* The infants and their parents/legally acceptable representative could comply with all of the scheduled visits in the study and the study requirements related to protocol compliance.
* The parents/legally acceptable representative (LAR) signed the written consent form.

Exclusion Criteria:

* Had previously received Haemophilus influenzae type b vaccine prior to this clinical study.
* Had a plan for vaccination with the vaccine other than those permitted in the protocol based on the standard vaccination schedule.
* Had been contacted with a patient with confirmed Hib infection within 30 days before the study start.
* Had had fever of ≥ 37.5°C within the last 3 days (If measured by tympanic thermometer, fever of 38°C or higher)
* Had or were suspected for immune function disorders; had previously received or were suspected to receive the immunosuppressive therapy; or had received the immunosuppressive therapy within 30 days prior to participating in the study (including systemic corticosteroids or inhalation corticosteroids) (However, it was not the exclusion criteria to have received corticosteroid therapy (prednisolone equivalent ≤ 0.5 mg/kg/day) not more than for 14 consecutive days at least 30 days before their participation in the study).
* Had received the treatment of parenteral immunoglobulin or blood products after birth.
* Had allergic history to be considered due to any component of the vaccine including excipients or preservatives.
* Three preceding generations in an ancestral line were not of Korean heritage.
* Had or were suspected to have significant disorders of blood, heart, liver, kidney, nervous system, respiratory system, or digestive system, or the investigator decided that the evaluation of study objective might be interrupted.
* Had been treated with other investigational drug by participating in another clinical trial within 30 days prior to this study entry, or were participating in another clinical study at that time.
* Had plans to move away from the area of the study site before completing the study.
* Inappropriate to take part in this clinical study in the principal investigator or sub-investigator's opinion, for the reasons other than above criteria.

Ages: 49 Days to 84 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 217 (Actual)
Dates: Start 2007-07; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have obtained protective antibody response with anti-PRP antibody titer not less than 1㎍/mL after the 3rd vaccination (at 4 weeks after the 3rd vaccination) in the test group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, Jongno-gu, South Korea

REFERENCES:
- [Derived] Kim KH, Kim YK, Kim NH, Chang SH, Lee J, Park EA, Park SE, Eun BW, Lee H, Lee HJ. Immunogenicity and safety of LBVH0101, a new Haemophilus influenzae type b tetanus toxoid conjugate vaccine, compared with Hiberix in Korean infants and children: a randomized trial. Vaccine. 2012 Feb 27;30(10):1886-94. doi: 10.1016/j.vaccine.2011.12.122. Epub 2012 Jan 13. PMID 22245607